CLINICAL TRIAL: NCT04757935
Title: The Effects of Yoga on Disease Activity in Youth With Inflammatory Bowel Disease: a Pilot Feasibility Study
Brief Title: Yoga for Youth With IBD: a Pilot Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB Protocol 37755
Record Dates: First submitted 2018-09-06; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases; Yoga; Adolescents; Crohn Disease; Ulcerative Colitis
Keywords: inflammatory bowel disease; adolescent; yoga; mind-body
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Yoga — Yoga for 30 minutes three times weekly for 8 weeks in addition to three, 1-hour in-studio yoga sessions.

SUMMARY:
An 8-week yoga intervention to determine the feasibility and acceptability of yoga as a supplemental therapy in the management of inflammatory bowel disease in the adolescent population.

DETAILED DESCRIPTION:
Youth with IBD experience abdominal pain, diarrhea, weight loss, and psychological suffering related to their disease process. While many biologic and non-biologic therapies are available to target the inflammatory component of IBD, youth with IBD could benefit from a more holistic therapy that addresses psychological wellness, which has been shown, in turn, to reduce disease burden. It is known that stress (multiple varieties) leads to IBD flares. It is also known that mind-body intervention reduces stress. The mind-gut connection is widely discussed in medical circles, however, current therapies have not capitalized on it. The investigators would like to know if an easily accessible mind-body intervention (yoga) can improve wellness, lower stress levels, and reduce intestinal inflammation in youth with IBD.

The study will be an 8-week feasibility pilot. Participants will be asked to participate in online yoga videos and in-studio yoga sessions. Participants will be asked to complete multiple surveys throughout the intervention and continue receiving standard care from their primary gastroenterology team.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-21
* Diagnosis of Crohn's Disease or Ulcerative Colitis
* Patient of a Stanford Children's Health or Stanford-affiliated Pediatric Gastroenterologist
* Ability to attend in-person meetings/training

Exclusion Criteria:

* Initiation of biologic therapy in prior 3 months
* Hospital admission in prior 2 months
* Major surgery in prior 1 month
* PUCAI/PCDAI >65
* Current pregnancy
* Severe developmental or intellectual disability
* Non-english speaking
* Not participating in another concurrent clinical trial

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of acceptability | 1 hour focus group at conclusion of intervention.
  Focus Group

SECONDARY OUTCOMES:
Fecal Calprotectin | 6 weeks (Prior to intervention; After conclusion of intervention)
  Stool biomarker that indicates intestinal inflammation
Pediatric Ulcerative Colitis Activity Index | 6 weeks (Prior to intervention; After conclusion of intervention)
  5 question assessment tool for disease tracking for patient's with ulcerative colitis
PROMIS-37 | 6 weeks (Prior to intervention; After conclusion of intervention)
  NIH Pediatric Assessment Tool

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ming Yeh, MD, Principal Investigator — Clinician Educator at Stanford University; Jenna Marie Arruda, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No